CLINICAL TRIAL: NCT00236509
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Response Study to Evaluate the Efficacy and Safety of Topiramate in the Prophylaxis of Migraine
Brief Title: A Study of the Efficacy and Safety of Topiramate in the Prevention of Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002254
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Migraine; Common Migraine; Classic Migraine; Headache
Keywords: Migraine; Common Migraine; Classic Migraine; Headache; Topiramate; Prophylaxis
MeSH Terms: conditions — Migraine Disorders; Migraine without Aura; Migraine with Aura; Headache | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of three doses of topiramate (50 milligrams[mg], 100mg, and 200mg taken daily) compared with placebo in the prevention of migraine.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, multi-center study to evaluate the effectiveness and safety of three different doses of topiramate (50mg, 100mg, and 200mg daily) in migraine prophylaxis. The study consists of five phases: baseline (determination of whether patients meet the eligibility criteria and tapering of any migraine medication patients are already taking); initial titration and double-blind phase (8 weeks) which begins with 25 mg/daily increasing to the assigned (50, 100, 200 mg/day topiramate); followed by a maintenance period at the target dose (18 weeks); tapering transition phase (up to 7 weeks); and open-label extension up to 6 months (to a maximum topiramate dose of 1600 mg/day); doses are adjusted to maximize effectiveness and minimize side effects. The primary study hypothesis is that one or more of the three doses of topiramate (50, 100, 200 mg/day) will be superior to placebo in the prophylaxis of migraine based on the change in monthly (28 day) migraine period rate from the prospective baseline period to the double-blind phase and that topiramate treatment is well tolerated. During the titration period (8 weeks), doses are increased to target dose of daily topiramate (50 milligrams[mg], 100, or 200mg) or placebo, taken twice daily by mouth. Doses are continued for 18 weeks, adjusted over 7 weeks, and continued for up to 6 months during the Open-Label Extension.

ELIGIBILITY:
Inclusion Criteria:

* Medical history consistent with migraine with or without aura according to the International Headache Society (IHS) for at least 6 months prior to the study
* Between 3 to 12 migraine periods and no greater than 15 headache days (migraine and non-migraine) per month during the Baseline Phase
* No clinically significant abnormalities on neurological exams, electrocardiogram (ECG) or clinical laboratory test results at baseline
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Patients with headaches other than migraine
* Patients with episodic tension or sinus headaches
* Onset of migraine after age of 50 years
* Patients who have failed more than two adequate regimens for migraine prophylaxis
* Patients who overuse pain medications or certain other medications

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 2001-02; Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Changes in length of time between the onset and cessation of painful migraine symptoms (migraine period) from the baseline. Safety evaluations conducted throughout the study.

SECONDARY OUTCOMES:
Proportion of patients responding to the treatment. Changes from baseline to double-blind phase in number of monthly migraine attacks, monthly migraine days, number of days/month requiring rescue medication, and Health-Related Quality of Life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Silberstein SD, Neto W, Schmitt J, Jacobs D; MIGR-001 Study Group. Topiramate in migraine prevention: results of a large controlled trial. Arch Neurol. 2004 Apr;61(4):490-5. doi: 10.1001/archneur.61.4.490. PMID 15096395